CLINICAL TRIAL: NCT01694498
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Trial Investigating the Efficacy and Safety of Two Different Dose Levels of Desmopressin for the Treatment of Nocturia in Adult Men
Brief Title: Comparative Trial to Investigate the Efficacy and Safety of Desmopressin for the Treatment of Nocturia in Adult Men
Acronym: NOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000030
Record Dates: First submitted 2012-09-11; First posted 2012-09-27 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A. Desmopressin 25 µg (Active Comparator): 1 orally disintegrating tablet every night during study period
  Interventions: Drug: A: Desmopressin 25 µg
- B. Desmopressin 50 µg (Active Comparator): 1 orally disintegrating tablet every night during study period
  Interventions: Drug: B. Desmopressin 50 µg
- C. Placebo (Placebo Comparator): 1 orally disintegrating tablet every night during study period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: A: Desmopressin 25 µg
  Arms: A. Desmopressin 25 µg
Drug: B. Desmopressin 50 µg
  Arms: B. Desmopressin 50 µg
Drug: Placebo
  Arms: C. Placebo

SUMMARY:
The purpose of the study is to investigate the efficacy and safety of two different dose levels of desmopressin orally disintegrating tablets against placebo for the treatment of nocturia in adult men during 12 weeks treatment

ELIGIBILITY:
Inclusion Criteria:

* Has given written consent prior to any trial-related activity is performed
* Male sex, aged 20 years or older
* At least 2 nocturnal voids every night in a consecutive 3-day period as documented in the diary during the screening period
* Has given agreement about contraception during the trial

Exclusion Criteria:

* Suspicion of bladder outlet obstruction or a urine flow of less than 5 mL/s as confirmed by uroflowmetry after suspicion of bladder outlet obstruction
* A surgical treatment for bladder outlet obstruction or prostatic hyperplasia within the past 6 months
* Showing symptoms of any of the following diseases: Benign prostatic obstruction; Interstitial cystitis; Overactive bladder, defined as >6 daytime voids, ≥1 urgency episode, and ≥1 urge urinary incontinence episode per 24 hours as documented in the 3-day diary period; Severe stress urinary incontinence
* Chronic prostatitis/chronic pelvic pain syndrome
* Psychogenic or habitual polydipsia
* Urinary retention or a post void residual volume in excess of 150 mL as confirmed by bladder ultrasound performed after suspicion of urinary retention
* Cancer
* A history of urologic malignancies or a history of cancer which has not been in remission for the last 5 years
* Genito-urinary tract pathology
* Neurogenic detrusor activity
* Suspicion or evidence of heart failure
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Hepatobiliary diseases: Aspartate aminotransferase >80 U/L or alanine aminotransferase >90 U/L; Total bilirubin >1.5 mg/dL
* Renal insufficiency: Serum creatinine level >1.09 mg/dL; Estimated glomerular filtration rate <50 mL/min
* Hyponatraemia: Serum sodium level <135 mEq/L
* Central or nephrogenic diabetes insipidus
* Syndrome of inappropriate antidiuretic hormone
* Obstructive sleep apnea
* Previous desmopressin treatment
* Treatment with another investigational product within the past 3 months
* Concomitant treatment with any prohibited medication
* Alcohol or substance abuse
* A job or lifestyle that may interfere with regular night-time sleep
* A mental condition, lack of decision-making ability, dementia, a speech handicap, or any other reason which, in the judgement of the investigator (sub-investigator), would impair the participation in the trial

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of nocturnal voids | During 12 weeks

SECONDARY OUTCOMES:
Change from baseline in mean time to first void | During 12 weeks
Responder status (33% reduction in nocturnal voids) | During 12 weeks
Change from baseline in mean number of nocturnal voids | 1, 4, 8 and 12 weeks
Change from baseline in mean time to first void | 1, 4, 8 and 12 weeks
Responder status (33% reduction in nocturnal voids) | 1, 4, 8 and 12 weeks
Change from baseline in mean nocturnal urine volume | 1, 4, 8 and 12 weeks
Change from baseline in nocturnal polyuria index | 1, 4, 8 and 12 weeks
Change from baseline in the effect on sleep disturbance | 1, 4, 8 and 12 weeks
Change from baseline in the impact on quality of life | 12 weeks
Adverse events, changes from baseline in serum sodium level, laboratory values | During 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (35):
- Japan (35):
  - Clinic Tsudanuma, Chiba
  - University of Fukui Hospital, Fukui
  - Kato Clinic, Gunma
  - Umeyama Clinic, Gunma
  - Harada Urology Clinic, Hyōgo
  - Sakaguchi Urological Clinic, Hyōgo
  - Nakamura Urology Clinic, Kanagawa
  - Nishi-Yokohama International Hospital, Kanagawa
  - Yokohama Shinmidori General Hospital, Kanagawa
  - Izumino Hospital, Bouchikai, Kochi
  - Kamei Clinic, Kochi
  - Den Urology Clinic, Osaka
  - Iwasa Clinic, Osaka
  - Kanno Clinic, Osaka
  - Morimoto Clinic, Osaka
  - Naka Clinic, Osaka
  - Uemura Clinic, Osaka
  - Urology department Kuroda Clinic, Osaka
  - Yamaguchi Clinic, Osaka
  - Yamanaka Clinic, Osaka
  - Fukuda Clinic, Saitama
  - Yasuda Urology Clinic, Saitama
  - Hirano Clinic, Tokyo
  - Hirata Internal Medicine Urology Clinic, Tokyo
  - J Tower Clinic, Tokyo
  - Koganeibashi Sakura Clinic, Tokyo
  - Kunitachi Sakura Hospital, Tokyo
  - Kusunoki Clinic, Tokyo
  - Moriguchi Clinic, Tokyo
  - Nakanoma Clinic Urology Department, Tokyo
  - Ogawa Clinic, Tokyo
  - Ogikubo Ekimae Clinic, Tokyo
  - Shibuya Shin-minamiguchi Clinic, Tokyo
  - Tokyo Kamata Hospital, Tokyo
  - Toru Clinic, Tokyo